CLINICAL TRIAL: NCT02586051
Title: A Phase Ib, Single- and Multiple-Dose, Open-Label Study of The Safety, Pharmacokinetics and Pharmacodynamics of Obinutuzumab in Adults With End-Stage Renal Disease and Hypersensitization Awaiting Renal Transplantation
Brief Title: A Study of Obinutuzumab to Evaluate Safety and Tolerability in Hypersensitized Adult Participants With End Stage Renal Disease Awaiting Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WT29749
Record Dates: First submitted 2015-10-23; First posted 2015-10-26 (Estimated); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Kidney Failure, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — obinutuzumab; Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes

ARMS (2):
- Cohort 1: Single Dose Obinutuzumab (Experimental): Desensitization period: Participants will receive obinutuzumab on Day 1 followed by high dose intravenous immunoglobulin (IVIG) on Days 22 and 43 of treatment period.
  Transplantation period: Participants who are found to qualify for transplantation and receive a compatible kidney offer after inclusion will receive two additional infusions of obinutuzumab (one at the time of transplantation [within the first 48 hours of the transplantation] and second at Week 24 post-transplantation).
  Interventions: Drug: Obinutuzumab; Drug: Intravenous Immunoglobulin
- Cohort 2: Repeated Dose Obinutuzumab (Experimental): Desensitization period: Participants will receive obinutuzumab on Days 1 and 15 followed by high dose IVIG on Days 22 and 43. An additional dose of obinutuzumab may be administered on Day 169 at investigator's discretion.
  Transplantation period: Participants who are found to qualify for transplantation and receive a compatible kidney offer after inclusion will receive two additional infusions of obinutuzumab (one at the time of transplantation [within the first 48 hours of the transplantation] and second at Week 24 post-transplantation).
  Interventions: Drug: Obinutuzumab; Drug: Intravenous Immunoglobulin

INTERVENTIONS:
Drug: Obinutuzumab — Obinutuzumab 1000 milligrams (mg) IV infusion.
  Other Names: RO5072759
Drug: Intravenous Immunoglobulin — High dose (2 grams per kilogram [g/kg]) IVIG (maximum 140 grams).

SUMMARY:
This is a Phase Ib, open-label study of single and repeat doses of obinutuzumab administered as intravenous (IV) infusion in adults with end stage renal disease (ESRD). Participants will be enrolled into two cohorts receiving either one (Cohort 1) or two or more (Cohort 2) obinutuzumab infusions. Both cohorts will receive standard pretreatments to reduce the risk of infusion-related reactions (IRRs).

Desensitization Period: In Cohort 1, participants will receive single dose obinutuzumab IV infusion on Day 1. Following review of Cohort 1 aggregated safety data up to 4 weeks post dose for the last participant of Cohort 1, Cohort 2 will be allowed to proceed. In Cohort 2, participants will receive obinutuzumab IV infusion on Days 1 and 15. Transplantation Period: Participants who qualify for transplantation and receive a compatible kidney offer after inclusion in Cohort 1 or Cohort 2 will receive two additional infusions (one at the time of transplantation and second at Week 24 post-transplantation) of obinutuzumab. Assessment of the safety and tolerability of the obinutuzumab regimen will be conducted at Week 24 of the desensitization phase and at Week 28 post-transplantation. All participants will be monitored for a minimum of 12 months following the last obinutuzumab infusion.

ELIGIBILITY:
Inclusion Criteria:

* ESRD with a history of sensitizing events
* United network for organ sharing (UNOS) listed for a deceased donor kidney transplantation
* Estimated high likelihood of receiving an offer in the coming 12-18 months from screening as evidenced by: present on at least one match run for a deceased donor kidney during the past year, or calculated panel reactive antibody (cPRA) greater than or equal to (≥) 98 percent (based on revisions to allocation policy introduced in 2014)
* Female participants of childbearing potential: agreement to remain abstinent or use two adequate methods of contraception during the treatment period and for at least 18 months after the last dose of study drug
* Male participants: agreement to remain abstinent or use contraceptive measures and agreement to refrain from donating sperm during the treatment period and for at least 12 months after the last dose of study drug

Exclusion Criteria:

* Incomplete recovery from recent major surgery or less than (<) 12 weeks since major surgery prior to baseline and participants planned surgery within 24 weeks of baseline except for kidney transplantation
* Pregnant or lactating women
* Positive serum human chorionic gonadotropin (hCG) measured at screening unless considered not clinically significant based on best medical judgement and if reassessment after ≥48 hours shows a less than a 2-fold rise from previous level
* Primary or secondary immunodeficiency disease
* Seropositivity for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) or seropositivity for Hepatitis C
* History of active or latent tuberculosis (TB) or suspicion of active TB
* Known active infection of any kind or any major episode of infection requiring hospitalization or treatment with IV anti-infective agents within 4 weeks of baseline or completion of oral anti-infective agents within 2 weeks prior to baseline
* Currently active alcohol or drug abuse or history of alcohol or drug abuse
* Participants with a history of prior kidney transplantation(s) after 6 participants with prior kidney transplants will be enrolled in the study
* Participants on peritoneal dialysis with a history of peritoneal infection at any time during the 12 weeks from prior to screening
* Participants on peritoneal dialysis with a positive culture or high cell count numbers on peritoneal fluid indicative of confirmed or suspected infection at the time of screening.
* Participants for synchronous organ transplant
* Recipients of any live attenuated vaccine(s) within 1 month of the screening visit
* Abnormal screening laboratory results
* Participants with a history of major cardiovascular or pulmonary disease
* Use of investigational agents within 12 weeks or five half-lives of randomization
* Use of an anti-CD20 therapy within the past 12 months
* Known contraindications to obinutuzumab
* History of severe allergic or anaphylactic reactions to monoclonal antibodies or components of obinutuzumab infusion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-11-19 (Actual); Primary Completion 2018-11-26 (Actual); Study Completion 2018-11-26 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events | Week 0 up to Week 24 of the desensitization phase

SECONDARY OUTCOMES:
Maximum Serum Concentration (Cmax) of Obinutuzumab During the Entire Study | Baseline up to last follow up (up to 76 weeks post-transplantation) (detailed timeframe is given in outcome measure description)
  Detailed timeframe:
  Cohort 1: Pre-dose (0 hour [hr]); within 1 hr of end of infusion; at 24 hr post-start of infusion at Day 1; Weeks 3 and 6 (immediately prior to IVIG administration); at Weeks 1, 2, 12, 24, 36 and 52; early termination and long-term follow up visit (up to Week 76).
  Cohort 2: Pre-dose (0 hr), within 1 hr of end of infusion, at 24 hr post-start of infusion at Week 0 and Week 2; immediately prior to IVIG administration at Week 3 and 6; Weeks 24 (pre-dose [0 hr] and within 1 hr of end of infusion if optional third infusion is provided); additionally at Weeks 1, 12, 36; and 52; at early termination and long-term follow-up visit (up to Week 76).
  Transplantation Period (Cohorts 1 and 2) (for participants undergoing transplantation): Pre-dose (0-30 minutes) and within 1 hr of end of infusion for each obinutuzumab dose at Weeks 0 and 24), at long-term follow-up visit (Week 76). Duration of infusion: approximately 4.5 hr for 1st infusion, and 3.5 hr for subsequent infusions.
Cmax of Obinutuzumab After the First Course of Obinutuzumab (Cmax1) | Baseline up to Week 2 (detailed timeframe is given in outcome measure description)
  Cohort 1: Pre-dose (0 hr); within 1 hr of the end of infusion; at 24 hr post-start of infusion at Day 1; at Weeks 1, 2 Cohort 2: Pre-dose (0 hr), within 1 hour of the end of infusion, at 24 hours post-start of infusion at Week 0; Pre-dose (0 hr) at Week 2 Duration of infusion: approximately 4.5 hr.
Cmax of Obinutuzumab After the Second Course of Obinutuzumab (Cmax2) | Cohort 2: Pre-dose (0 hr), within 1 hour of the end of infusion, at 24 hours post-start of infusion at Week 2 Duration of infusion: approximately 3.5 hr.
Area Under the Concentration Time Curve (AUC) of Obinutuzumab | Baseline up to last follow up (up to 76 weeks post-transplantation) (detailed timeframe is given in outcome measure description)
  Detailed timeframe:
  Cohort 1: Pre-dose (0 hr); within 1 hr of end of infusion; at 24 hr post-start of infusion at Day 1; Weeks 3 and 6 (immediately prior to IVIG administration); at Weeks 1, 2, 12, 24, 36 and 52; early termination and long-term follow up visit (up to Week 76).
  Cohort 2: Pre-dose (0 hr), within 1 hr of end of infusion, at 24 hr post-start of infusion at Week 0 and Week 2; immediately prior to IVIG administration at Week 3 and 6; Weeks 24 (pre-dose [0 hr] and within 1 hr of end of infusion if optional third infusion is provided); additionally at Weeks 1, 12, 36; and 52; at early termination and long-term follow-up visit (up to Week 76).
  Transplantation Period (Cohorts 1 and 2) (for participants undergoing transplantation): Pre-dose (0-30 minutes) and within 1 hr of end of infusion for each obinutuzumab dose at Weeks 0 and 24), at long-term follow-up visit (Week 76). Duration of infusion: approximately 4.5 hr for 1st infusion, and 3.5 hr for subsequent infusions.
Systemic Clearance (CL) of Obinutuzumab | Baseline up to last follow up (up to 76 weeks post-transplantation) (detailed timeframe is given in outcome measure description)
  Detailed timeframe:
  Cohort 1: Pre-dose (0 hr); within 1 hr of end of infusion; at 24 hr post-start of infusion at Day 1; Weeks 3 and 6 (immediately prior to IVIG administration); at Weeks 1, 2, 12, 24, 36 and 52; early termination and long-term follow up visit (up to Week 76).
  Cohort 2: Pre-dose (0 hr), within 1 hr of end of infusion, at 24 hr post-start of infusion at Week 0 and Week 2; immediately prior to IVIG administration at Week 3 and 6; Weeks 24 (pre-dose [0 hr] and within 1 hr of end of infusion if optional third infusion is provided); additionally at Weeks 1, 12, 36; and 52; at early termination and long-term follow-up visit (up to Week 76).
  Transplantation Period (Cohorts 1 and 2) (for participants undergoing transplantation): Pre-dose (0-30 minutes) and within 1 hr of end of infusion for each obinutuzumab dose at Weeks 0 and 24), at long-term follow-up visit (Week 76). Duration of infusion: approximately 4.5 hr for 1st infusion, and 3.5 hr for subsequent infusions.
Volume of Distribution at Steady State (Vss) of Obinutuzumab | Baseline up to last follow up (up to 76 weeks post-transplantation) (detailed timeframe is given in outcome measure description)
  Detailed timeframe:
  Cohort 1: Pre-dose (0 hr); within 1 hr of end of infusion; at 24 hr post-start of infusion at Day 1; Weeks 3 and 6 (immediately prior to IVIG administration); at Weeks 1, 2, 12, 24, 36 and 52; early termination and long-term follow up visit (up to Week 76).
  Cohort 2: Pre-dose (0 hr), within 1 hr of end of infusion, at 24 hr post-start of infusion at Week 0 and Week 2; immediately prior to IVIG administration at Week 3 and 6; Weeks 24 (pre-dose [0 hr] and within 1 hr of end of infusion if optional third infusion is provided); additionally at Weeks 1, 12, 36; and 52; at early termination and long-term follow-up visit (up to Week 76).
  Transplantation Period (Cohorts 1 and 2) (for participants undergoing transplantation): Pre-dose (0-30 minutes) and within 1 hr of end of infusion for each obinutuzumab dose at Weeks 0 and 24), at long-term follow-up visit (Week 76). Duration of infusion: approximately 4.5 hr for 1st infusion, and 3.5 hr for subsequent infusions.
Half-life (t1/2) of Obinutuzumab | Baseline up to last follow up (up to 76 weeks post-transplantation) (detailed timeframe is given in outcome measure description)
  Detailed timeframe:
  Cohort 1: Pre-dose (0 hr); within 1 hr of end of infusion; at 24 hr post-start of infusion at Day 1; Weeks 3 and 6 (immediately prior to IVIG administration); at Weeks 1, 2, 12, 24, 36 and 52; early termination and long-term follow up visit (up to Week 76).
  Cohort 2: Pre-dose (0 hr), within 1 hr of end of infusion, at 24 hr post-start of infusion at Week 0 and Week 2; immediately prior to IVIG administration at Week 3 and 6; Weeks 24 (pre-dose [0 hr] and within 1 hr of end of infusion if optional third infusion is provided); additionally at Weeks 1, 12, 36; and 52; at early termination and long-term follow-up visit (up to Week 76).
  Transplantation Period (Cohorts 1 and 2) (for participants undergoing transplantation): Pre-dose (0-30 minutes) and within 1 hr of end of infusion for each obinutuzumab dose at Weeks 0 and 24), at long-term follow-up visit (Week 76). Duration of infusion: approximately 4.5 hr for 1st infusion, and 3.5 hr for subsequent infusions.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (9):
- United States (9):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UCSF, San Francisco, California
  - Stanford Health Care, Stanford, California
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Mayo Clinic - Minnesota, Rochester, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - The Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati College of Medicine, Cincinnati, Ohio
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Derived] Redfield RR, Jordan SC, Busque S, Vincenti F, Woodle ES, Desai N, Reed EF, Tremblay S, Zachary AA, Vo AA, Formica R, Schindler T, Tran H, Looney C, Jamois C, Green C, Morimoto A, Rajwanshi R, Schroeder A, Cascino MD, Brunetta P, Borie D. Safety, pharmacokinetics, and pharmacodynamic activity of obinutuzumab, a type 2 anti-CD20 monoclonal antibody for the desensitization of candidates for renal transplant. Am J Transplant. 2019 Nov;19(11):3035-3045. doi: 10.1111/ajt.15514. Epub 2019 Jul 23. PMID 31257724